CLINICAL TRIAL: NCT02330250
Title: Effectiveness of Pharmaceutical Care in the Adherence of Systemic Lupus Erythematosus Treatment in Rio de Janeiro: a Randomized Clinical Trial
Brief Title: Effectiveness of Pharmaceutical Care in the Adherence of Systemic Lupus Erythematosus Treatment
Acronym: ADELES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Hospital Universitario Pedro Ernesto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ADELES/002
Record Dates: First submitted 2014-12-30; First posted 2015-01-01 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Systemic Lupus Erythematosus; Medication Adherence
Keywords: Systemic Lupus Erythematosus; Pharmaceutical care; Pharmaceutical services; Medication adherence
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Medication Adherence | interventions — Pharmaceutical Services

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmaceutical Care (Experimental): The patients will receive guidance from a pharmacist based on the Dader Method for Pharmaceutical Care, in addition to the medical care habitually delivered by the hospital.
  Interventions: Other: Pharmaceutical Care
- Control (Sham Comparator): The control group will receive the medical care habitually provided by the hospital, and the follow-up by a non-pharmacist professional.
  Interventions: Other: Control

INTERVENTIONS:
Other: Pharmaceutical Care — The patients assigned for the intervention group will receive guidance from a pharmacist ("pharmaceutical consultation") in addition to the medical care habitually delivered by the hospital.
  The pharmacist will review the drug therapy, identifying current and potential problems related to the drug prescription, making a systematic assessment of the need, effectiveness and safety of all medications and their adequacy to the patient's life routine. A care plan will then be designed along with the patient that may include interventions and/or referral to other practitioners.
  Other Names: Pharmaceutical Services
  Arms: Pharmaceutical Care
Other: Control — The patients assigned to the control group will receive the medical care habitually provided by the hospital and will be attended by a non-pharmacist professional, who will provide hygiene/nutritional counseling and risk reduction, such as smoking cessation advice; use of estrogen-based contraceptive drugs; exposure to sunlight, proper use of sunscreen and clothes; nutritional guidance on the intake of low saturated-fat food. As usual, information about the use of medication will be provided by the attending physician.
  Arms: Control

SUMMARY:
This project aims to improve adherence rate through pharmaceutical care in patients with systemic lupus erythematosus (SLE) to help achieving therapeutic goals and finally to improve the quality of life of these patients.

DETAILED DESCRIPTION:
Adherence to treatment is a primary determinant for the effectiveness of health care. Non-compliance may lead to therapeutic failure, make more difficult and complex the management of chronic diseases or cause death. The effectiveness of interventions on adherence has an important impact in the health of the population. Systemic lupus erythematosus (SLE) is an autoimmune disease with high proportion of hospital admissions and deaths and high cost of treatment. The prevalence of adherence in this group of patients in Brazil is very low (31.7%) and the drug treatment is complex. Our aim is to assess the effectiveness of Pharmaceutical Care in the adherence of drug treatment by SLE patients attended in a Rheumatology outpatient clinic in Rio de Janeiro, Brazil.

Randomized clinical trial (pragmatic trial), in which 120 adult patients with confirmed SLE diagnosis will be followed for 12 months, and randomized in two groups: the intervention group (attended by a pharmacist according to the Dader Method for Pharmaceutical Care), and the control group (attended by a non-pharmacist professional with counseling on hygiene/nutrition and reduction of risks in lupus therapy). The main outcome will be adherence to drug therapy and secondary outcomes the improvement of the medical condition and the quality of life of the patients.

ELIGIBILITY:
Inclusion criteria:

* SLE diagnosis according to the 2012 SLICC (Systemic Lupus International Collaborating Clinics Group) SLE classification criteria.
* Treatment with corticosteroids and antimalarials.
* History of biopsy-proven lupus nephritis classes III, IV, or V (2003 International Society of Nephrology / Renal Pathology Society) or nephritic/nephrotic lupus flare not undergone to kidney biopsy.

Exclusion Criteria:

* Current renal replacement therapy.
* Renal transplantation.
* Ongoing pulse therapy with cyclophosphamide and/or methylprednisolone.
* Aid by caregiver.
* Any psychiatric illness.
* Inability to understand the questions of the questionnaire.
* Patients'unwillingness to sign the informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2014-07; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 12 months
  Medication adherence will be measured by use of the eight-item Morisk Medication Adherence Scale (MMAS) translated and validated to brazilian portuguese

SECONDARY OUTCOMES:
SLE disease activity | 12 months
  SLE disease activity measured by use of Safety of Estrogens in Systemic Lupus National SLE Assessment Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI)
Quality of life | 12 months
  Quality of life measured by use of Medical Outcomes Study 36 - Item Short-Form Health Survey)

CONTACTS AND LOCATIONS:
Overall Officials: Jose FS Verani, PhD, Study Chair — Oswaldo Cruz Foundation
Locations (1):
- Reumathology outpatient clinics Pedro Ernesto University Hospital, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] de Oliveira-Filho AD, Morisky DE, Neves SJ, Costa FA, de Lyra DP Jr. The 8-item Morisky Medication Adherence Scale: validation of a Brazilian-Portuguese version in hypertensive adults. Res Social Adm Pharm. 2014 May-Jun;10(3):554-61. doi: 10.1016/j.sapharm.2013.10.006. Epub 2013 Oct 26. PMID 24268603
- [Background] Silva C, Canhao H, Barcelos A, Miranda L, Pinto P, Santos MJ. [Protocol for evaluation and monitoring of Systemic Lupus Erythematosus (PAMLES)]. Acta Reumatol Port. 2008 Apr-Jun;33(2):210-8. Portuguese. PMID 18604187
- [Background] Campolina AG, Ciconelli RM. [SF-36 and the development of new assessment tools for quality of life]. Acta Reumatol Port. 2008 Apr-Jun;33(2):127-33. Portuguese. PMID 18604180
- [Background] Oliveira-Santos M, Verani JF, Klumb EM, Albuquerque EM. Evaluation of adherence to drug treatment in patients with systemic lupus erythematosus in Brazil. Lupus. 2011 Mar;20(3):320-9. doi: 10.1177/0961203310383736. Epub 2010 Dec 23. PMID 21183558
- [Background] Barber N, Parsons J, Clifford S, Darracott R, Horne R. Patients' problems with new medication for chronic conditions. Qual Saf Health Care. 2004 Jun;13(3):172-5. doi: 10.1136/qhc.13.3.172. PMID 15175485
- [Background] Petri M, Orbai AM, Alarcon GS, Gordon C, Merrill JT, Fortin PR, Bruce IN, Isenberg D, Wallace DJ, Nived O, Sturfelt G, Ramsey-Goldman R, Bae SC, Hanly JG, Sanchez-Guerrero J, Clarke A, Aranow C, Manzi S, Urowitz M, Gladman D, Kalunian K, Costner M, Werth VP, Zoma A, Bernatsky S, Ruiz-Irastorza G, Khamashta MA, Jacobsen S, Buyon JP, Maddison P, Dooley MA, van Vollenhoven RF, Ginzler E, Stoll T, Peschken C, Jorizzo JL, Callen JP, Lim SS, Fessler BJ, Inanc M, Kamen DL, Rahman A, Steinsson K, Franks AG Jr, Sigler L, Hameed S, Fang H, Pham N, Brey R, Weisman MH, McGwin G Jr, Magder LS. Derivation and validation of the Systemic Lupus International Collaborating Clinics classification criteria for systemic lupus erythematosus. Arthritis Rheum. 2012 Aug;64(8):2677-86. doi: 10.1002/art.34473. PMID 22553077
- [Derived] Oliveira-Santos M, Verani JF, Camacho LA, de Andrade CA, Ferrante-Silva R, Klumb EM. Effectiveness of pharmaceutical care for drug treatment adherence in patients with systemic lupus erythematosus in Rio de Janeiro, Brazil: study protocol for a randomized controlled trial. Trials. 2016 Apr 2;17:181. doi: 10.1186/s13063-016-1317-1. PMID 27038611
- See also: Método Dáder. Guía de Seguimiento Farmacoterapêutico — http://www.pharmanet.com.br/atencao/metododader.pdf